CLINICAL TRIAL: NCT06788639
Title: Non-interventional Cohort Study of Patients Treated With Liso-cel (Lisocabtagene Maraleucel) for Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma in the Post-Marketing Setting
Brief Title: A Study of Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma Treated With Lisocabtagene Maraleucel in the Post-Marketing Setting
Status: Recruiting | Type: Observational
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CA082-1092
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants treated with lisocabtagene maraleucel
  Interventions: Biological: Lisocabtagene maraleucel

INTERVENTIONS:
Biological: Lisocabtagene maraleucel — According to the United States Prescribing Information

SUMMARY:
The purpose of this study is to characterize the long-term safety of lisocabtagene maraleucel (liso-cel), focusing on patients treated in the chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) indication, and will be part of post-marketing liso-cel pharmacovigilance activities

ELIGIBILITY:
Inclusion Criteria:

• Participants must have been treated in the post-marketing setting with ≥1 infusion of lisocabtagene maraleucel used for the treatment of relapsed/refractory (R/R) chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) within the approved indication and dosage per the United States Prescribing Information (USPI) and product specifications approved for commercial release in the USA

Exclusion Criteria:

* Participants known to be participating in investigational studies at the time of lisocabtagene maraleucel infusion
* Patients treated with non-conforming CAR T-cell product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults with relapsed/refractory chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) that are being treated with lisocabtagene maraleucel and are registered within the Center for International Blood and Marrow Transplant Research (CIBMTR) registry.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2044-06-30 (Estimated); Study Completion 2044-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to 15 years

SECONDARY OUTCOMES:
Complete remission rate (CRR | Up to 15 years
Overall response rate (ORR) | Up to 15 years
Progression-free survival (PFS) | Up to 15 years
Overall survival (OS) | Up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Center for International Blood and Marrow Transplant Research (CIBMTR), Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts